CLINICAL TRIAL: NCT04773574
Title: Physiologic Ocular Changes During Pregnancy in Women With High Myopia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Suthasinee Sinawat, Associate Professor, Khon Kaen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HE631583
Record Dates: First submitted 2021-02-25; First posted 2021-02-26 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: High Myopia; Pregnancy Related
Keywords: high myopia; pregnancy; choroidal thickness; retinal vascular density; retinal nerve fiber layer thickness; corneal curvature
MeSH Terms: interventions — Corneal Topography; Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal pregnant women with high myopia (Experimental): Corneal topography, Optical coherence tomography (OCT) and Optical coherence tomography angiography (OCTA) were performed in each trimesters and at 6 weeks after childbirth.
  Interventions: Device: Corneal topography, Optical coherence tomography (OCT) and Optical coherence tomography angiography (OCTA)

INTERVENTIONS:
Device: Corneal topography, Optical coherence tomography (OCT) and Optical coherence tomography angiography (OCTA) — Ocular investigations were performed in each trimesters and at 6 weeks after childbirth.
  1. st trimester : gestational age 8-12 weeks
  2. nd trimester : gestational age 24-28 weeks
  3. rd trimester : gestational age 34-38 weeks

SUMMARY:
The prevalence of myopia is seemingly increasing, and it is one of the major causes of blindness. High myopia is defined as a refractive error with spherical equivalent exceeding -6 diopters and/or the axial length longer than 26.5 mm. The global prevalence of high myopia is estimated to rise from 2.7% of the world population in 2010 to 9.8% of the world population in 2050. High myopia is characterized by axial length elongation, and consequent stretching of the posterior eye wall (thin retina and choroid). There are many complications of high myopia such as posterior staphyloma, lacquer cracks and myopic choroidal neovascularization. Normal labour may cause the ocular complication in pregnant women with high myopia, such as macular hemorrhage. Therefore, the caesarean section with epidural anesthesia is recommended. Moreover, there is no standard screening guideline for pregnant women with high myopia.

DETAILED DESCRIPTION:
There are few studies of posterior ocular changes during pregnancy. A recent meta-analysis showed that the choroidal thickness and retinal vascular density were increased during pregnancy especially in the 3rd trimester. From the literature review, there is only one publication of physiologic ocular changes during pregnancy in high myopia. Chen et al demonstrated that the choroidal thickness was increased significantly in the 3rd trimester. However, the changes of retinal vascular density in pregnant women with high myopia have never been studied before.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* high myopia: spherical equivalent > 6 diopters and/or axial length > 26.5 mm
* singleton pregnancy
* clear ocular media
* written inform consent

Exclusion Criteria:

* high risk pregnancy such as pre-eclampsia, gestational diabetes mellitus, hyperthyroidism and asthma.
* history of retinal diseases such as macular edema and retinal vascular occlusion
* history of intraocular inflammation or endophthalmitis
* history of intraocular laser treatment
* history of intraocular surgery

Withdrawal criteria

* childbirth before 34 weeks' gestation
* multifetal pregnancy was detected by ultrasound
* high risk pregnancy which could not follow the research protocol such as severe pre-eclampsia
* retinal diseases occur during the follow-up period such as central serous chorioretinopathy, retinal detachment and choroidal neovascularization
* significant ocular trauma during the follow-up period
* severe peripartum or postpartum complications such as thromboembolic disease and postpartum hemorrhage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Choroidal thickness | 40 weeks
  Choroidal thickness was measured by optical coherence tomography

SECONDARY OUTCOMES:
Retinal vascular density | 40 weeks
  Percentage of retinal vascular density was measured by optical coherence tomography angiography
Retinal nerve fiber layer thickness | 40 weeks
  Retinal nerve fiber layer thickness was measured by optical coherence tomography
Corneal thickness | 40 weeks
  Corneal thickness was measured by corneal topography
Corneal curvature | 40 weeks
  Corneal curvature was measured by corneal topography

CONTACTS AND LOCATIONS:
Overall Officials: Suthasinee Sinawat, MD, Principal Investigator — KKU Eye Center, Department of Ophthalmology, Faculty of Medicine, Khon Kaen University

IPD SHARING:
Plan to Share IPD: No